CLINICAL TRIAL: NCT02555241
Title: Instructional Programming to Promote the Emergence of Generative Language in Children With Autism Spectrum Disorder
Brief Title: Emergence of Generative Language
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Alice Shillingsburg, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00080641
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD, Children
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- One Baseline Session (Experimental): Designated for participants #1 and #2. Participants complete 1 Baseline Session followed immediately by 12 weeks of standard treatment. Standard treatment will require the participant to attend clinic-based treatment sessions for 1 hour per day, 3 days per week, for 12 weeks. Standard treatment will consist of 3 components: mand training, matrix training, and stimulus equivalence training.
  Interventions: Behavioral: Mand Training; Behavioral: Matrix; Behavioral: Stimulus Equivalence Training
- Two Baseline Sessions (Experimental): Designated for participants #3 and #4. Participants complete a Baseline Session followed by a 12 week wait period before repeating a Baseline Session followed immediately by 12 weeks of standard treatment. Standard treatment will require the participant to attend clinic-based treatment sessions for 1 hour per day, 3 days per week, for 12 weeks. Standard treatment will consist of 3 components: mand training, matrix training, and stimulus equivalence training.
  Interventions: Behavioral: Mand Training; Behavioral: Matrix; Behavioral: Stimulus Equivalence Training
- Three Baseline Sessions (Experimental): Designated for participants #5 and #6. Participants complete a Baseline Session followed by two repetitions of the Baseline Session (each 12 weeks apart) and 12 weeks of standard treatment immediately following the third session. Standard treatment will require the participant to attend clinic-based treatment sessions for 1 hour per day, 3 days per week, for 12 weeks. Standard treatment will consist of 3 components: mand training, matrix training, and stimulus equivalence training.
  Interventions: Behavioral: Mand Training; Behavioral: Matrix; Behavioral: Stimulus Equivalence Training

INTERVENTIONS:
Behavioral: Mand Training — The mand training component of treatment will consist of behavioral principles designed to increase the participant's Mean Length of Utterances (MLU) when manding.
Behavioral: Matrix — The matrix training component of treatment will consist of behavioral principles designed to teach labeling of noun-verb and color-shape combinations using matrix training.
Behavioral: Stimulus Equivalence Training — The stimulus equivalence training component of treatment is designed to examine the emergence of untrained skills following the training of relational skills.

SUMMARY:
The purpose of this study is to investigate the effects of several applied behavior teaching procedures on the use of multi-word utterances by children with autism.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder (ASD)
* Provide a diagnostic report confirming a diagnosis of ASD and/or obtain a total raw score of 15 or greater on the Social Questionnaire Lifetime Form (SCQ)
* Speaks primarily in one word utterances
* English as their primary language
* Follows simple 1-step instructions
* Transportation/availability to attend 3, 1-hour sessions each week for 12 weeks

Exclusion Criteria:

* Children with significant problem behavior that interferes with structured intervention

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2015-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in Mean Length of Utterances (MLU) during manding | Baseline (Up to 24 Weeks), End of Standard Treatment (Up to 36 weeks)
  The mean length of utterances (MLU) during manding will be evaluated in a 10 minute probe. The goal of intervention is to increase of MLU to an average of 3 words per mand.
Acquisition of noun-verb and color-shape combinations during tacting | Baseline (Up to 24 Weeks), End of Standard Treatment (Up to 36 weeks)
  The goal of intervention is mastery of 80% of evaluated noun-verb and color-shape targets.
Emergence of intraverbal responses | Baseline (Up to 24 Weeks), End of Standard Treatment (Up to 36 weeks)
  The goal of intervention is the mastery of 80% of evaluated intraverbal responses (2 for each target, 18 total).

SECONDARY OUTCOMES:
Change in Macarthur Bates-Communicative Development Inventory (CDI) Score | Baseline (Up to 24 Weeks), End of Standard Treatment (Up to 36 weeks)
  The Macarthur Bates-Communicative Development Inventory (CDI) is completed by a parent/caregiver and evaluates current word use . A higher score indicates the use of more words.
Observe overall improvements in pragmatic language within social/play interactions with parents/caregivers, as measured on the Direct Observation of Spoken Language (DOSL). | Baseline (Up to 24 Weeks), End of Standard Treatment (Up to 36 weeks)
  A goal of the intervention is to observe an increase in spontaneous mands, an increase in spontaneous tacts, as well as an increase in intraverbal responses.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Shillingsburg, Principal Investigator — Emory University Assistant Professor